CLINICAL TRIAL: NCT00246207
Title: An Open-label Study Evaluating the Safety and Effectiveness of OROS Methylphenidate Hydrochloride (CONCERTA) in Adults With Attention Deficit Hyperactivity Disorder
Brief Title: CONCERTA (OROS Methylphenidate Hydrochloride) for the Treatment of Attention Deficit Hyperactivity Disorder in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003097
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; once-day oral tablets
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: CONCERTA (OROS methylphenidate hydrochloride)

SUMMARY:
The purpose of this pilot study is to evaluate the safety, tolerability and potential effectiveness of CONCERTAÂ® (methylphenidate hydrochloride extended-release tablets), a central nervous system (CNS) stimulant for the treatment of adults with Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
CONCERTA® is a long-acting form of methylphenidate (a CNS stimulant). Methylphenidate is a recognized first-line treatment for ADHD in children and adolescents. It is widely acknowledged in the scientific literature that the disorder often will persist in adulthood, and is associated with significant morbidity and undesirable outcomes. Despite this, few studies have been conducted to investigate the efficacy and safety of stimulant therapy in treating ADHD in adults. As a consequence, drug treatment options for adult sufferers of ADHD are limited. The primary objective of this pilot, open-label study is to evaluate the safety, tolerability and potential effectiveness of CONCERTA® (18, 36, 54 or 72 mg of methylphenidate hydrochloride, administered once-daily) in adult subjects with Attention Deficit Hyperactivity Disorder (ADHD). Patients cannot have been treated with any methylphenidate- or amphetamine-containing medication within 4 weeks of screening visit. Once deemed eligible, subjects will be started on 18 mg of CONCERTA® once-daily for 3 days, titrated up on Day 4 to 36 mg and maintained at this dose for 7 days. Depending on patient response, the dose of CONCERTA® can continue to be titrated up every 7 days, first to 54 mg and then to a maximum of 72 mg per day, in order to achieve the optimal dose for each patient. The primary efficacy outcomes will be the changes from baseline to the end of treatment in the inattention and hyperactivity/impulsivity subscale scores of the investigator-rated Conners' Adult ADHD Rating Scale (CARRS). Safety and tolerability will be monitored throughout the study. The study hypothesis is that stimulant therapy in treating adult ADHD will be safe and effective, measured by the Conners' Adult ADHD Rating Scale (CAARS) score. CONCERTA® is taken orally, once-daily. Starting with CONCERTA® 18 mg for 3 days, subjects are titrated up on Day 4 to 36 mg for 7 days. Depending on response, tolerability and clinician's discretion, the dose of CONCERTA® can continue to be titrated up every 7 days, first to 54 mg and then to a maximum of 72 mg per day (two 36 mg tablets), until each subject's optimal dose is achieved. The titration period will last a maximum of 24 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Attention Deficit Hyperactivity Disorder (ADHD) according to the Diagnostic and Statistical Manual of Mental Diseases (DSM-IV) obtained via clinical interview and confirmed by the Wender Utah Rating Scale
* ADHD symptoms from childhood to adulthood, with some symptoms present before age 7 years which continue to meet DSM-IV criteria at the time of assessment. (ADHD is not diagnosed if the symptoms are better accounted for by another psychiatric disorder.)
* investigator-rated CAARS (Conners' Adult ADHD Rating Scale) baseline score greater than or equal to 24
* Clinical Global Impression of Severity baseline score greater than or equal to 4 and a total Montgomery Asberg Depression Rating score at baseline of less than or equal to 16.

Exclusion Criteria:

* Have been treated with any methylphenidate- or amphetamine-containing medication within 4 weeks of screening visit
* any clinically unstable psychiatric condition including the following, but not limited to: acute mood disorder, schizophrenia, bipolar disorder, acute obsessive compulsive disorder, anti-social personality disorder
* subjects with marked anxiety, tension, aggression or agitation, Autism or Asperger's syndrome
* a diagnosis of substance abuse or dependence within 6 months prior to screening evaluation
* use of other psychotropic medications used to treat non-ADHD psychiatric disorders, if the dose of the medication has not remained stable for a minimum of 4 weeks prior to trial entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-03; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness outcomes will be the changes in the inattention and hyperactivity/impulsivity subscale scores of the investigator-rated CAARS (Conners' Adult ADHD Rating Scale) from baseline to the end of treatment.

SECONDARY OUTCOMES:
The changes in other effectiveness assessments will be secondary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Result] Fallu A, Richard C, Prinzo R, Binder C. Does OROS-methylphenidate improve core symptoms and deficits in executive function? Results of an open-label trial in adults with attention deficit hyperactivity disorder. Curr Med Res Opin. 2006 Dec;22(12):2557-66. doi: 10.1185/030079906X154132. PMID 17166338
- See also: An open-label study evaluating the safety and effectiveness of OROS* Methylphenidate (CONCERTA*) in adults with Attention Deficit Hyperactivity Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=357&filename=CR003097_CSR.pdf